CLINICAL TRIAL: NCT03241849
Title: New Surgical Technique To Control Postpartum Hemorrhage Due To Placenta Accreta
Brief Title: Surgical Technique To Control Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STPPGE
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified surgical technique for placenta accreta (Other)
  Interventions: Procedure: Modified surgical technique for placenta accreta

INTERVENTIONS:
Procedure: Modified surgical technique for placenta accreta — suturing of the myometrium splitted by the placenta in cases presented by placenta accreta

SUMMARY:
Placenta accreta is an obstetrical complication where the placenta becomes firmly adherent to the uterine wall. Placenta accreta can lead to considerable maternal morbidity and mortality due to hemorrhage, infection, or other surgical complications such as those resulting from hysterectomy. Retained placenta accreta is usually a rare condition, but its prevalence is increasing due to the rise in the rate of deliveries by Cesarean section.

Placenta accreta is a potentially life-threatening obstetric condition that requires a multidisciplinary approach to management. The incidence of placenta accreta has increased and seems to parallel the increasing cesarean delivery rate. Women at greatest risk of placenta accreta are those who have myometrial damage caused by a previous cesarean delivery with either an anterior or posterior placenta previa overlying the uterine scar. Diagnosis of placenta accreta before delivery allows multidisciplinary planning in an attempt to minimize potential maternal or neonatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated gestational age between 34 -40 weeks .
2. Presence of total or focal parts of placenta accreta "morbidly adherent placenta" .
3. Cases with mild vaginal bleeding or not having any vaginal bleeding

Exclusion Criteria:

1. Severe attack of bleeding require an immediate intervention.
2. Associated with placental abruption
3. Patients with known bleeding disorders or on anticoagulant therapy.
4. Preoperative decision to do peripartum hysterectomy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss (mL) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided